CLINICAL TRIAL: NCT03509727
Title: Point-of-care-testing for Procalcitonin in Diagnosis of Bacterial Infections in Young Infants: a Diagnostic Accuracy Study
Brief Title: Procalcitonin in Diagnosis of Bacterial Infections in Young Infants
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Thomas Waterfield, Dr Thomas Waterfield, Belfast Health and Social Care Trust
Other Study IDs: PCT
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A diagnostic accuracy study investigating the accuracy of procalcitonin in diagnosing invasive bacterial infections in your infants.

DETAILED DESCRIPTION:
The primary aim of this study was to report on the diagnostic accuracy of procalcitonin in the diagnosis of bacterial infections in young infants. This included invasive bacterial infections; defined as the isolation of a bacterial pathogen in blood or cerebrospinal fluid culture.

We conducted a prospective observational diagnostic accuracy study. Young infants less than 90 days of age presenting to the Royal Belfast Hospital for Sick Children with signs of possible bacterial infection were eligible for inclusion. Eligible infants underwent procalcitonin testing using 0.5ml of whole blood with a BRAHMS assay on the Samsung LABGEO IB10® analyser.

ELIGIBILITY:
Inclusion Criteria:

* Suspected bacterial infection

Exclusion Criteria:

* None

Max Age: 90 Days | Sex: All
Age Groups: Child
Study Population: All young infants presenting to the emergency department with suspected infection are eligible for testing.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Invasive bacterial infection | 2 days
  Isolation of a bacterial pathogen in blood or cerebrospinal fluid culture

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shields, Principal Investigator — Queen's University, Belfast
Locations (1):
- Royal Belfast Hopsital for Sick Children, Belfast, United Kingdom

REFERENCES:
- [Derived] Waterfield T, Maney JA, Hanna M, Fairley D, Shields MD. Point-of-care testing for procalcitonin in identifying bacterial infections in young infants: a diagnostic accuracy study. BMC Pediatr. 2018 Dec 12;18(1):387. doi: 10.1186/s12887-018-1349-7. PMID 30541505